CLINICAL TRIAL: NCT07292506
Title: The Impact of Acupuncture on Biomarkers of Brain Injury and Inflammatory Response in Migraine
Acronym: ACUPMIGRAINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-319/2024-2711-6
Record Dates: First submitted 2025-11-18; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Migraine; Migraine Headache; Migraine Headache, With or Without Aura; Migraine in Adults
Keywords: electroacupuncture; migraine; acupuncture; biomarkers of brain injury; inflammatory response; laser acupuncture; traditional acupuncture
MeSH Terms: conditions — Migraine Disorders | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Participants will be randomly placed into one of three groups:
  Traditional Acupuncture - standard acupuncture treatment on local scalp and distal points Electroacupuncture - standard acupuncture on local scalp points combined with gentle electrical stimulation of the needles placed on distal points Laser Acupuncture - standard acupuncture on local scalp points combined with low-level laser instead of needles on distal acupuncture points
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard acupuncture (Active Comparator): Traditional Acupuncture - standard acupuncture treatment on local scalp and distal points
  Interventions: Other: Standard acupuncture
- Electroacupuncture (Active Comparator): Electroacupuncture - standard acupuncture on local scalp points combined with gentle electrical stimulation of the needles placed on distal points
  Interventions: Other: Standard acupuncture; Other: Electroacupuncture
- Laser Acupuncture (Active Comparator): Laser Acupuncture - standard acupuncture on local scalp points combined with low-level laser instead of needles on distal acupuncture points
  Interventions: Other: Standard acupuncture; Other: Laser Acupuncture

INTERVENTIONS:
Other: Standard acupuncture — standard acupuncture on the scalp and distal acupuncture point that will not be stimulated with electro or laser device
Other: Electroacupuncture — Electroacupuncture - distal acupuncture points will be stimulated will electronic device that is used for electroacupuncture
  Arms: Electroacupuncture
Other: Laser Acupuncture — Distal acupuncture points will be stimulated with laser needles
  Arms: Laser Acupuncture

SUMMARY:
Migraine is more than just a headache-it can involve changes in the brain and inflammation. Recent research suggests that acupuncture may help by calming pain signals and reducing inflammation in the body. Scientists are studying whether acupuncture can also lower certain markers in the blood that show brain stress or inflammation. While more research is needed, acupuncture is considered safe and may reduce the number and severity of migraine attacks for many people. Acupuncture has been used for over 40 years in our practice to manage acute and chronic pain, including migraines. When performed by trained physicians, it is safe and typically reduces headache frequency and intensity, as well as nausea and vomiting, lowering the need for pain medication.

Investigators are exploring three different ways to help manage migraine headaches using gentle stimulation techniques. These include laser acupuncture, electroacupuncture, and traditional acupuncture.

Investigators want to see which method works best for reducing migraine symptoms. Investigators will look at how participants feel after treatment and also check blood samples for signs of inflammation and certain substances linked to migraines, such as calcitonin gene-related peptide (CGRP) and markers of brain stress.

Investigators have a goal to find safe and effective options that can improve migraine care and help people feel better.

DETAILED DESCRIPTION:
Investigators are conducting a study to compare three different types of acupuncture treatments. Each participant will be carefully evaluated to meet the requirements for participation. Before joining, each participant will have a conversation with investigators to explain the study and answer any questions.

Participants will be randomly placed into one of three groups:

Traditional Acupuncture - standard acupuncture treatment Electroacupuncture - standard acupuncture combined with gentle electrical stimulation.

Laser Acupuncture - standard acupuncture combined with acupuncture using a low-level laser instead of needles.

After the treatment, Investigators will check in with participants again after 1 and 3 months to see how they are feeling and whether the effects have lasted.Participation is voluntary, with no financial compensation, and care will not be affected by the decision to participate.

Outcomes will be assessed using questionnaires before treatment and for three months afterward, measuring migraine days, pain intensity, medication use, headache frequency, and satisfaction of participants. Blood samples will be collected at baseline, after treatment, and three months later to analyze migraine-related biomarkers. Results will be statistically evaluated. Investigators expect acupuncture to reduce headache severity and medication use.

So far, there has been no direct comparison of these three methods. Investigators want to find out:

Which method works best. How long the benefits last. Whether participants need repeat treatments.

ELIGIBILITY:
Inclusion Criteria

* Adults diagnosed with migraine headaches according to the International Classification of Headache Disorders (ICHD).
* Patients who are not currently receiving monoclonal antibodies targeting CGRP (Calcitonin Gene-Related Peptide)
* Ability to provide informed consent and comply with study procedures. Exclusion Criteria
* Use of CGRP monoclonal antibody therapy within the past 6 months.
* Other significant neurological or systemic conditions that could interfere with study outcomes.
* Pregnancy or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
NRS 3 | Baseline and three months from last acupuncture stimulation
  Pain intensity three months after treatment measured with NRS (Numeric rate scale) from 0 (for = pain) to 10 (maximal pain)

SECONDARY OUTCOMES:
HIT- 6 | Baseline and three months from last acupuncture stimulation
  HIT-6 stands for Headache Impact Test - 6 items.Higher scores indicate a greater impact of migraine on the life of partcipants. The four headache impact severity categories are little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78) Score range 36-78 It is widely used for people with migraine or other headache disorders. The goal is to understand the impact of headaches on daily functioning, not just pain intensity.
MIDAS | Baseline and three months from last acupuncture stimulation
  The MIDAS questionnaire stands for Migraine Disability Assessment. It is a tool used to measure how much migraines affect a person's daily life and productivity. Scores on the MIDAS are highly correlated with physician judgments about the severity of illness and need for treatment. The score of this instrument is as follows: little or no disability, 5 to 10; moderate disability, 1 to 20; and severe disability, more than 20.
Biomarkers of brain injury and inflammatory response | Baseline, day of last acupuncture stimulation and three months from last acupuncture stimulation
  We will take blood samples for interleukin - 6, 8 and 10 (Il6, IL8, IL10), leptin, Nerve growth factor (NGF), S100 calcium-binding protein A8 (S100A8), Brain-derived neurotrophic factor (BDNF) and CGRP

CONTACTS AND LOCATIONS:
Overall Officials: Lea Rupert, MD, Principal Investigator — Clinical department of anaesthesiology and surgical intensive therapy University Medical Centre Ljubljana; Jasmina Markovic Bozic, MD, Phd, Asist. Prof., Study Chair — Clinical department of anaesthesiology and surgical intensive therapy University Medical Centre Ljubljana
Locations (1):
- Clinical department of anaesthesiology and surgical intensive therapy University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu S, Yu L, Luo X, Wang M, Chen G, Zhang Q, Liu W, Zhou Z, Song J, Jing H, Huang G, Liang F, Wang H, Wang W. Manual acupuncture versus sham acupuncture and usual care for prophylaxis of episodic migraine without aura: multicentre, randomised clinical trial. BMJ. 2020 Mar 25;368:m697. doi: 10.1136/bmj.m697. PMID 32213509
- [Result] Liu Y, Yu S. Recent Approaches and Development of Acupuncture on Chronic Daily Headache. Curr Pain Headache Rep. 2016 Jan;20(1):4. doi: 10.1007/s11916-015-0535-7. PMID 26700695
- [Result] Peters GL. Migraine overview and summary of current and emerging treatment options. Am J Manag Care. 2019 Jan;25(2 Suppl):S23-S34. PMID 30681821